CLINICAL TRIAL: NCT04066621
Title: Efficacy and Safety of CRO-SBT Performed in Children With Acute Bacterial Infection
Brief Title: PHase IV Clinical Trial of Ceftriaxone Sodium and Sulbactam Sodium for Injection (CRO-SBT)
Acronym: CRO-SBT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiangbei Welman Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LENVOCRO (2012)CSSSI-0.4
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Respiratory Tract Infections; Urinary Tract Infections in Children
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Ceftriaxone; Sulbactam; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRO-SBT (Experimental): Ceftriaxone Sodium and Sulbactam Sodium for Injection(2:1)
  Interventions: Drug: Ceftriaxone Sodium and Sulbactam Sodium for Injection

INTERVENTIONS:
Drug: Ceftriaxone Sodium and Sulbactam Sodium for Injection — daily dose was 75 mg/kg by weight, 1-2 times ivgtt per day, 4 to 14 days
  Other Names: weipufen

SUMMARY:
To evaluate the safety and efficacy of treatment of children with acute bacterial infection disease with Ceftriaxone Sodium and Sulbactam Sodium for Injection in the condition of widely used, and provide the basis of adjusting the dosage regimen for children in particular.

DETAILED DESCRIPTION:
Ceftriaxone sodium and sulbactam sodium for injection (2:1)plays a therapeutic role by the former inhibiting bacterial cell wall synthesis，the latter making irreversible competitive inhibition of β-lactamase.The antimicrobial effect of Ceftriaxone can be enhanced by the two combined. The compound specifically aims to the mechanism of bacterial resistance, extending the life of Ceftriaxone in the treatment-resistant pathogen infections.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children ages≥6 years to< 14 years.
* Weight≥18kg who in hospital or outpatients with good compliance;
* The subjects were diagnosed as respiratory infection, urinary tract infection or other infection caused by the compound sensitive bacteria after clinical symptoms and signs laboratory examination and auxiliary examination according to the clinically recognized diagnostic criteria, and should be treated with systemic antibiotics;
* Subjects had not used effective antimicrobial agents before screening, or had used antimicrobial agents but the efficacy was not obvious;
* No severe liver and kidney cardiovascular and hematopoietic diseases were found in the subjects (AST and ALT were not more than 1.5 times of the upper limit of normal value,Cr was within the normal range);
* Subject guardian informed consent and/or subject's own informed consent subject volunteers to participate in this study and has signed the subject's informed consent.

Exclusion Criteria:

* History of hypersensitivity reactions to carbapenems, cephalosporins, penicillin, other β-lactam antibiotics;
* Patients with specific infections who require treatment with other antimicrobial agents;
* Use of penicillin roxithromycin vitamin B vitamin C and other drugs may interfere with the efficacy or safety evaluation of drugs at the same time;
* Patients at risk of serious drug interactions due to combination of medications;
* Patients who have other diseases and thought to affect efficacy evaluations or be poor compliance;
* Attended clinical trial in three monthes.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-06-11 (Actual); Study Completion 2017-05-27 (Actual)

PRIMARY OUTCOMES:
The cure rate of patients | Seven days after treatment
  Clinically effective/Clinically ineffective

SECONDARY OUTCOMES:
bacterial clearance rate | 48 hours after treatment
  end of treatment of bacteriological efficacy (bacterial clearance rate)

CONTACTS AND LOCATIONS:
Overall Officials: yuhua hu, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No